CLINICAL TRIAL: NCT01378312
Title: A Phase I Randomized Placebo-Controlled, Double-Blind Study to Evaluate Safety and Immunogenicity of AERAS-402 When Administered to HIV-Negative BCG-Vaccinated Adults Without Evidence of Tuberculosis Infection
Brief Title: A Study to Evaluate Safety and Immunogenicity of AERAS-402
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-004-402
Record Dates: First submitted 2011-02-24; First posted 2011-06-22 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2012-11

CONDITIONS: Tuberculosis
Keywords: vaccine; TB; tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Arm (Placebo Comparator)
  Interventions: Biological: Placebo
- AERAS 402 Arm (Active Comparator)
  Interventions: Biological: AERAS 402

INTERVENTIONS:
Biological: AERAS 402 — 0.5 mL IM injection of 3 x 1010vp AERAS-402 on Study Days 0 and 28
  Arms: AERAS 402 Arm
Biological: Placebo — 0.5 mL IM injection of 0vp (Placebo) on Study Days 0 and 28
  Arms: Placebo Arm

SUMMARY:
This Phase I study will be conducted as a randomized, double-blind, placebo-controlled study in healthy adult subjects who are HIV-negative, BCG-vaccinated, and have no evidence of tuberculosis infection. The study will be conducted at one clinical research site in India.

The available live tuberculosis vaccine, Bacillus Calmette-Guérin (BCG), provides incomplete protection against pulmonary tuberculosis. For unknown reasons, a BCG revaccination or "booster", while not toxic, does not provide much additional protection. AERAS-402 presents tuberculosis antigens in the setting of a new, live, replication-deficient adenovirus vaccine that may increase T cell-mediated immunity and thus protection from tuberculosis. Since BCG-vaccinated individuals are the population for which AERAS-402 might be indicated, AERAS-402 will be administered to individuals already vaccinated with BCG.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female
* Is age 18 through 45 years on Study Day 0
* Has completed written informed consent
* Had BCG vaccination at least 5 years ago, documented through medical history or presence of scar
* Has general good health, confirmed by medical history and physical examination
* Has Body Mass Index (BMI) between 19 and 30 (kg/m2)
* Has ability to complete follow-up period of 182 days as required by the protocol
* Females: Ability to avoid pregnancy from 28-days prior to initial study vaccination through the duration of their participation in the study.
* Will commit to avoiding elective surgery for the duration of the study
* Has ability to stay in contact with the investigative site for the duration of the study
* Has completed simultaneous enrollment in Aeras Vaccine Development Registry protocol

Exclusion Criteria:

* Acute illness on the day of randomization
* Oral temperature ≥37.5°C on the day of randomization
* Evidence of significant active infection
* Used immunosuppressive medication within 42 days before entry into the study
* Received immunoglobulin or blood products within 42 days
* Received any investigational drug therapy or vaccine within 182 days
* Received any standard vaccine within 42 days
* Participated in any clinical trial of an investigational adenovirus-based vaccine previously.
* Current chronic drug therapy
* History or laboratory evidence of any past, present or future possible immunodeficiency state which will include (but is not limited to) any laboratory indication of HIV infection
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine
* Previous medical history that may compromise the safety of the subject in the study
* Evidence of a new acute illness that may compromise the safety of the subject in the study
* Evidence of chronic hepatitis (e.g., hepatitis B core antibody, or hepatitis C antibody, or other)
* Inability to discontinue daily medications except contraceptives during the study period
* History of alcohol or drug abuse within the past 2 years
* Tobacco or cannabis smoking three or more days per week
* Positive urine test for illicit drugs (opiates, cocaine, amphetamines)
* History or evidence of any systemic disease on physical examination
* History or evidence (including chest X-ray) of active tuberculosis
* Shared a residence within the last year with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis
* All females: Positive urine pregnancy test during screening; positive serum pregnancy test on the day of study vaccination; are nursing
* Abnormal (per local laboratory parameters) hemoglobin, hematocrit, white blood cell count, absolute neutrophil count, absolute lymphocyte count, prothrombin time (PT), partial thromboplastin time (PTT), serum creatinine, GGT, ALT, AST, total bilirubin, alkaline phosphatase (ALP), or creatinine drawn within 36 hours prior to randomization.
* Laboratory test evidence of Mtb infection
* Tuberculin skin test evidence of Mtb infection, defined as 15 mm of induration or greater.
* Anal intercourse with another man at least one time (with or without condoms)
* Exchange of goods, money, services or drugs for sex.
* Use of intravenous drugs.
* Sexual intercourse or genital contact within the last 12 months with a known HIV positive individual
* Vaginal intercourse within the last 12 months without use of a condom with a known user of intravenous drugs
* Oral to genital contact within the last 12 months with a known user of intravenous drug
* Vaginal intercourse within the last 12 months without use of a condom with an individual known to have more than one sex partner
* Oral to genital contact within the last 12 months with an individual known to have more than one sex partner

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number and Percentage of Adverse Events by treatment group | Day 56
  The number and percentage of Adverse Events will be presented and compared by treatment group (placebo vs AERAS 402).

SECONDARY OUTCOMES:
Immune Response | Day 182
  Percentage of CD4 and CD8 cells producing specific cytokines will be measured and tabulated in subjects who have received the vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Vanya Dhagat, MD, Principal Investigator — Lotus Labs
Locations (1):
- Lotus Labs, Bangalore, Bangalore, India

REFERENCES:
- [Derived] Hoft DF, Blazevic A, Stanley J, Landry B, Sizemore D, Kpamegan E, Gearhart J, Scott A, Kik S, Pau MG, Goudsmit J, McClain JB, Sadoff J. A recombinant adenovirus expressing immunodominant TB antigens can significantly enhance BCG-induced human immunity. Vaccine. 2012 Mar 9;30(12):2098-108. doi: 10.1016/j.vaccine.2012.01.048. Epub 2012 Jan 30. PMID 22296955